CLINICAL TRIAL: NCT04209387
Title: Neurophysiology Markers of PTSD's Presence, Severity and Therapy Outcome
Brief Title: Novel EEG Coherence Biomarkers for PTSD Assessment
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: D2846-R
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PTSD Undergoing Psycho-therapy: Veterans with PTSD seeking treatment and undergoing psycho-therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy to Improve Social Support for Veterans with PTSD ( ACT-SS)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy to Improve Social Support for Veterans with PTSD ( ACT-SS) — ACT is an evidence-based treatment that focuses on identifying a person's valued life goals and explicitly targets experiential avoidance to assist clients in committing to behavior change aligned with their values and becoming more psychologically flexible

SUMMARY:
Current practice for diagnosing and managing PTSD relies primarily on subjective clinical assessments by clinicians as well as patient self-report. An independent, objective and neuro-physiology based method for directly assessing brain function is not available, but is much needed to improve diagnosis and management of PTSD. To address this critical need, the investigators propose to test a set of novel biomarkers which are based on measures of coherent activity among the regions of cerebral cortex during sleep. In preliminary studies on EEG acquired during sleep from Veterans with PTSD alone as well as other co-morbidities, the investigators have shown that the neuromarkers were highly sensitive/specific to the presence of PTSD, and highly sensitive to the severity of symptoms in PTSD group. The overall goal of this project is to further validate these novel neurophysiology marker in retrospective and prospective studies

DETAILED DESCRIPTION:
This is a prospective study with PTSD (n=50) at multiple times during the Veterans ongoing clinical treatment for PTSD. Sleep EEG measures will be collected at pretreatment, after first session of therapy, immediately after completion of therapy, and at 3-month post therapy.

Methodology:

N=50 Veterans with PTSD symptoms undergoing the Veterans clinical treatment at the Bedford VA will be recruited and the following data will be acquired: Sleep-EEG, Demographic, Medical History, and Use of Medications forms, The Beck Depression Inventory, Pittsburgh Sleep Quality Index, Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form, NIH PROMIS, PCL-5, and Clinician-Administered PTSD Scale (CAPS-5). Primary independent variable will be changes in the Neuromarker and the dependent variables will consist of the functional and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who have been previously deployed and meet diagnostic criteria for PTSD. Prior traumatic experience(s) does not have to be direct combat (e.g. may include search and rescue of combat operations). Persons previously treated for PTSD will be eligible so long as current diagnostic criteria are present. Specific inclusion criteria are as follows:

  * Current (past month) diagnosis of PTSD as determined from the 30-item CAPS (score >45).
  * History of deployment and combat-related exposure stated as the principal reason for seeking treatment (based on self-report).
  * Ability to read and speak English to complete surveys and participate in therapy.
  * Explicit denial of suicidal or homicidal ideation or intent, which will be corroborated by reviewing the patient chart.

Exclusion Criteria:

* Brain injury prohibiting speech, writing, and purposeful actions.
* Identified to have current suicidal or homicidal ideation (immediate referral to a crisis center/hospital).
* Major confounding psychiatric disorder; i.e. assessment indicates presence of:

  * Major mental health disorder that involves psychosis
  * Otherwise in the state of psychological crisis (appropriate referral to occur)
  * Current or recent (within 1 month of study entry) DSM-5 substance use disorder
  * Individuals who are taking either illicit or prescribed Rx that could interfere with EEG, including benzodiazepines and certain mood stabilizers (e.g., Lithium)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans who have been previously deployed and meet diagnostic criteria for PTSD. Prior traumatic experience(s) does not have to be direct combat (e.g. may include search and rescue of combat operations). Persons previously treated for PTSD will be eligible so long as current diagnostic criteria are present.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mo Modarres, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modarres M, Cochran D, Kennedy DN, Frazier JA. Comparison of comprehensive quantitative EEG metrics between typically developing boys and girls in resting state eyes-open and eyes-closed conditions. Front Hum Neurosci. 2023 Nov 6;17:1237651. doi: 10.3389/fnhum.2023.1237651. eCollection 2023. PMID 38021243

RESULTS

PARTICIPANT FLOW:
Groups:
- Veterans With PTSD Undergoing Therapy: Veterans with PTSD diagnosis undergoing psychotherapy tested at 3 time points, (1) before initiation of therapy, (2) at the end of therapy, (3) 3-months follow-up
Period: Overall Study
Arm/Group | Veterans With PTSD Undergoing Therapy
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Veterans With PTSD Undergoing Therapy: PTSD undergoing therapy to be studies before and after treatment
Arm/Group | Veterans With PTSD Undergoing Therapy
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 11
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 26
Coherence [Mean (Standard Deviation); unit: Coherence] | 0.28 (0.02)

OUTCOME MEASURES:

1. Primary Outcome: Coherence
Description: Coherence describes the degree of electrical activity (EEG) synchrony among brain regions. Coherence is equivalent to correlation coefficient in frequency domain and takes values from 0 (no synchrony) to 1 (perfect synchrony). A detailed description of this method is provided in: Modarres M, Cochran D, Kennedy DN, Frazier JA. Comparison of comprehensive quantitative EEG metrics between typically developing boys and girls in resting state eyes-open and eyes-closed conditions.
Time Frame: Pre-treatment (within one week of initiation of PTSD therapy), within one week before initiation of their treatment protocol, within one week after the conclusion of their treatment phase, and about three months after their last therapy session
Measure: Mean (Standard Deviation); unit: Coherence
Groups:
- PTSD Veterans Undergoing Psychotherap: Baseline (Before initiation of therapy)
Arm/Group | PTSD Veterans Undergoing Psychotherap
Number analyzed (Participants) | 26
Coherence
  Baseline (Before Initiation of Therapy | 0.28 (0.02)
  End ot Therapy | 0.27 (0.02)
  3-Month Follow-up | 0.27 (0.27)
Statistical Analysis 1: Comparison: PTSD Veterans Undergoing Psychotherap; Pair-wise comparison of changes in coherency from baseline (before therapy) to the end of therapy. Pair-wise comparison of changes in coherency from end of therapy to 3-month follow-up; Test type: Other — p < .01; p = 0.01, Wilcoxon (Mann-Whitney) — p adjusted for multiple comparisons; ANOVA test of means

ADVERSE EVENTS:
Time Frame: 6 months
Description: No Difference in Adverse Event Reporting
Groups:
- Veterans With PTSD Undergoing Psychotherapy: PTSD Veterans with PTSD diagnosis undergoing psycho-therapy tested at 3 time points, (1) before initiation of therapy, (2) at the end of therapy, (3) 3-months follow-up
Arm/Group | Veterans With PTSD Undergoing Psychotherapy
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04209387/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT04209387/ICF_001.pdf